CLINICAL TRIAL: NCT01370083
Title: Tongue Pressure Profile Training for Dysphagia Post Stroke
Acronym: TPPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Responsible Party: Principal Investigator, Catriona M. Steele, Senior Scientist, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRI-SRRL-0411-TPPT
Record Dates: First submitted 2011-06-03; First posted 2011-06-09 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Dysphagia
Keywords: Dysphagia; Viscosity; Tongue; Pressure
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stroke: TPPT (Experimental): Adults with dysphagia post stroke (within 4-16 weeks of onset) who have radiographically confirmed difficulties with thin liquid bolus control. Individuals will complete 24 sessions of tongue-pressure-profile training over 8-12 weeks.
  Interventions: Behavioral: Tongue Pressure Profile Training
- Stroke: TPSAT Control (Active Comparator): Individuals with dysphagia (within 4-16 weeks post stroke) who demonstrate difficulties with thin liquid control on videofluoroscopy. Individuals will complete 24 sessions of tongue-pressure strength-and-accuracy training over 8-12 weeks.
  Interventions: Behavioral: Tongue-Pressure Strength-and-Accuracy Training

INTERVENTIONS:
Behavioral: Tongue Pressure Profile Training — 60 tongue-pressure tasks per session, emphasizing control of the slope of tongue pressure release, informed by biofeedback. Pressures will be measured using a hand-held oral manometer (Iowa Oral Performance Instrument) with signals displayed on a computer.
  Other Names: Iowa Oral Performance Instrument
  Arms: Stroke: TPPT
Behavioral: Tongue-Pressure Strength-and-Accuracy Training — 60 tongue-pressure tasks per session, emphasizing maximum effort strength tasks and accuracy targets within 20-95% of each patient's maximum, informed by biofeedback. Pressures will be measured using a hand-held oral manometer (Iowa Oral Performance Instrument) with amplitude output in kiloPascals displayed on an LCD screen.
  Other Names: Iowa Oral Performance Instrument
  Arms: Stroke: TPSAT Control

SUMMARY:
People with swallowing impairment experience particular difficulty swallowing thin liquids safely; the fast flow of liquids makes them difficult to control. The tongue plays a critical role in containing liquids in the mouth, channeling the direction of their flow towards the pharynx (throat) and controlling their flow along that channel. The investigators are engaged in a program of research to better understand tongue function in swallowing, particularly with respect to controlling the flow of liquids. In this study the investigators will compare two different tongue-pressure resistance training protocols, to determine whether a protocol that emphasizes strength-and-accuracy or one that emphasizes pressure timing work better for improving liquid flow control in swallowing.

DETAILED DESCRIPTION:
Drinking thin liquids is something that most of us take for granted; yet this task is one that many patients with dysphagia (swallowing impairment) cannot do safely. Instead, these individuals receive liquids in thickened form: thickened juice, thickened coffee… even thickened water. The literature tells us that patients dislike the taste and feel of thickened liquids and find that their thirst is not quenched. Patients on thickened liquids are prone to inadequate fluid intake and dehydration. Many patients are non- compliant and drink thin liquids, despite documented risk for aspiration (i.e., airway invasion) and its consequences. Given these limitations, it is important that dysphagia researchers continue to pursue treatments with the potential to restore safe and functional thin liquid swallowing in people with dysphagia.

In the past decade, tongue pressure resistance training has emerged as an innovative treatment for dysphagia. Dr. JoAnne Robbins (University of Wisconsin - Madison)has shown that 8-weeks of intensive tongue pressure resistance training improves tongue strength in healthy seniors and those with dysphagia following stroke. In our lab (the Swallowing Rehabilitation Research Laboratory at the Toronto Rehabilitation Institute), the investigators have studied a variation on Dr. Robbins' treatment called "Tongue Pressure Strength and Accuracy Training". This approach also improves tongue strength and improves aspiration. However, the investigators continue to be bothered by the fact that people with dysphagia post stroke often have difficulty controlling the flow of thin liquids, even after these strength-focused protocols of tongue-pressure training.

The investigators have recently completed a study of tongue pressures profiles (strength and timing) in healthy people, which shows that tongue pressures are released more slowly with thin liquids than with thick liquids. This reveals active control of thin liquid flow, and suggests that both the strength and timing of tongue pressure play a role in flow-control. The investigators believe that treatment outcomes may be better if tongue pressure resistance training protocols take both strength and timing into consideration. To this end, the investigators have recently identified a subset of tongue pressure training tasks for which the strength and timing profile of tongue pressure onset and release is similar to that seen in liquid swallowing. The investigators propose that a treatment protocol will have better potential to yield favourable outcomes for thin liquid flow-control if it focuses on such tasks.

In this study, the investigators want to determine whether tongue pressure profile training, which addresses both timing and amplitude issues in tongue pressure generation, yields better functional outcomes in swallowing than strength-and-accuracy focused treatment. The investigators will pursue this question in a small randomized prospective trial, building on our prior work in this area.

The investigators will recruit 60 new patients with who demonstrate thin liquid flow-control difficulties secondary to stroke. These individuals will be randomized either to tongue-pressure strength-and-accuracy training (TPSAT) or to the novel intervention, tongue-pressure profile training (TPPT). The investigators will study their treatment outcomes after 12 weeks (24-sessions) of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with dysphagia characterized by prolonged swallow response duration for 5 cc boluses of thin liquid (i.e., > 350 ms, confirmed in videofluoroscopy).

Exclusion Criteria:

* premorbid reported history of swallowing, motor speech, gastro-esophageal or neurological difficulties.
* prior history of surgery to the speech apparatus (other than routine tonsillectomy or adenoidectomy).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catriona M Steele, Ph.D., Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Rehabilitation Institute - University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Steele CM, Bayley MA, Peladeau-Pigeon M, Stokely SL. Tongue pressure profile training for dysphagia post stroke (TPPT): study protocol for an exploratory randomized controlled trial. Trials. 2013 May 7;14:126. doi: 10.1186/1745-6215-14-126. PMID 23782628

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stroke: TPPT | Stroke: TPSAT Control
Started | 7 | 7
Completed | 5 | 6
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Individuals with dysphagia following stroke (within 4-16 weeks post onset) with radiographically confirmed difficulties with thin liquid bolus control.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stroke: TPPT | Stroke: TPSAT Control | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Full Range); unit: years] | 75 [56 to 84] | 67 [49 to 89] | 71 [49 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 7 | 14
Tongue Strength, Continuous [Mean (Standard Deviation); unit: Kilopascals] — 1 Repetition Maximum Isometric Tongue-Palate Pressure measured across 3 repetitions of maximum isometric tongue pressure generation using the Iowa Oral Performance Instrument, with the bulb located in a posterior position in the mouth (with the flat edge of the bulb aligned with the first molar tooth).
  Kilopascals | 12.71 (7.48) | 25.71 (8.36) | 19 (10)
Swallow Response Time (thin liquids), Categorical [Number; unit: participants] — This is a categorical measure (within vs.above normal limits) of the time interval between a thin liquid bolus entering the pharynx (passing the shadow of the ramus of mandible) and onset of upward-anterior hyolaryngeal excursion for the swallow. The continuous parameter is measured in milliseconds from videofluoroscopy. Durations < 350 ms are considered within normal limits; those > 350 ms are considered prolonged. Prolonged swallow response time on thin liquid swallows at baseline was an inclusion criterion for this study. We report the # of participants with values > 350 ms.
  participants | 7 | 7 | 14
Penetration-Aspiration, Categorical [Number; unit: participants] — The 8-point Penetration-Aspiration Scale is an ordinal rating scale used to rate the severity of airway invasion during swallowing. Scores of 1 and 2 are considered normal. Here we report the number of participants displaying abnormal scores (i.e. of 3 and higher) vs normal scores (1 or 2) on thin liquid swallows in videofluoroscopy.
  participants
    Abnormal Scores (3 or higher) | 4 | 4 | 8
    Normal Scores (1 or 2) | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Swallow Response Time for 5 cc Thin Liquid Swallows
Description: Swallow response time (the time duration between bolus passing the ramus of the shadow of the mandible and onset of hyolaryngeal excursion for airway protection 5cc thin liquid barium boluses in videofluoroscopy. Measures > 350 ms are considered to reflect impairment and a heightened risk of penetration-aspiration. The participant's mean swallow response time will be calculated across a series of 3 X 5 cc swallows and then reduced to a binary score < vs > 350 milliseconds.
Time Frame: Post treatment (12 weeks)
Measure: Number; unit: participants
Arm/Group | Stroke: TPPT | Stroke: TPSAT Control
Number analyzed (Participants) | 6 | 5
participants
  Number with values < 350 ms | 2 | 2
  Number with values > 350 ms | 4 | 3

2. Secondary Outcome: Penetration-Aspiration Scale Score for 5 cc Thin Liquid Swallows
Description: The Penetration-Aspiration Scale is an 8-point ordinal scale that addresses the depth of airway invasion and response to airway invasion during swallowing. We will measure penetration-aspiration for a series of 3 X 5 cc thin liquid swallows in videofluoroscopy. The participant's worst score will be taken to reflect their swallowing safety. This score will be collapsed into a binary score < vs. > 3 on the scale, reflecting material entering and remaining in or below the supraglottic space (versus transient entry or no entry at all).
Time Frame: Post-treatment (12 weeks)
Population: Participants with complete pre and post-treatment videofluoroscopy data available.
Measure: Number; unit: participants
Arm/Group | Stroke: TPPT | Stroke: TPSAT Control
Number analyzed (Participants) | 6 | 5
participants
  Swallowing safety within normal limits (scores <3) | 2 | 4
  Swallowing safety impaired (scores >2) | 4 | 1

3. Secondary Outcome: Tongue-palate Pressure Amplitude for Maximum Isometric Pressures
Description: We will measure the amplitude of peak tongue-pressure amplitudes on maximum isometric pressure tasks performed using the Iowa Oral Performance Instrument. The maximum amplitude across a series of 3 maximum isometric pressure tasks performed with the bulb in a posterior position (flat end aligned with the first molar tooth) will be used to document tongue strength.
Time Frame: Post-treatment value
Population: Individuals with complete pre and post-treatment data available
Measure: Mean (Standard Deviation); unit: Kilopascals
Arm/Group | Stroke: TPPT | Stroke: TPSAT Control
Number analyzed (Participants) | 6 | 5
Kilopascals | 28.45 (18.03) | 43.84 (13.33)

ADVERSE EVENTS:
Time Frame: During the 3 months of active participation in the study
Arm/Group | Stroke: TPPT | Stroke: TPSAT Control
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stroke: TPPT (N=7) | Stroke: TPSAT Control (N=7)
New Stroke Requiring Acute Care Hospitalization (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No